CLINICAL TRIAL: NCT02851056
Title: Evaluating the Safety and Biological Activity of a Dendritic Cell Survivin Vaccine in Patients With Multiple Myeloma Undergoing Autologous Hematopoietic Cell Transplantation
Brief Title: Survivin Vaccine : Multiple Myeloma Autologous Hematopoietic Cell Transplant (HCT)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18346
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Vaccine; Dendritic cell; autologous hematopoietic cell transplant; HCT
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — 13-valent pneumococcal vaccine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Survivin Vaccine and Autologous HCT (Experimental): Dendritic Cell Survivin Vaccine (DC:AdmS) and Autologous Hematopoietic Cell Transplantation (HCT). Participants will receive 1 pre-transplant survivin vaccine, 7-30 days prior to stem cell apheresis collection. After the first survivin vaccination, participants will be mobilized with Granulocyte-colony Stimulating Factor (G-CSF). A second survivin vaccine will be administered on day +21 (between day+20 and +34) after HCT. All participants will be co-immunized with Prevnar 13 at each time they receive the survivin vaccine.
  Interventions: Biological: Survivin Vaccine; Procedure: Autologous Hematopoietic Cell Transplantation; Biological: Prevnar 13; Drug: Granulocyte-colony Stimulating Factor

INTERVENTIONS:
Biological: Survivin Vaccine — Pre-transplant vaccination : The target dose of Survivin+ Dendritic cells (survivin+, CD11c+, Human Leukocyte Antigen - antigen D Related (HLA-DR)+ by flow-cytometry) is 15 x 10^6 cells. A minimum of 1 x 10^6 cells and a maximum of 20 x 10^6 cells will be administered.
  Post-transplant vaccination: The target dose of Survivin+ Dendritic cells (survivin+, CD11c+, HLA-DR+ by flow-cytometry) is 15 x 10^6 cells. A minimum of 1 x 10^6 cells and a maximum of 20 x 10^6 cells will be administered.
Procedure: Autologous Hematopoietic Cell Transplantation — The participant's own cells are collected from their blood, frozen, and then given back to them after they receive chemotherapy.
  Other Names: HCT
Biological: Prevnar 13 — 13-Valent Pneumococcal Conjugate Vaccine (PCV13, Prevnar13). Co-Immunization: All participants will be co-immunized with Prevnar at each time they receive the survivin vaccine. This vaccine will be administered intramuscular (IM) 0.5cc.
  Other Names: PCV13
Drug: Granulocyte-colony Stimulating Factor — After the first survivin vaccination, participants will be mobilized with G-CSF.
  Other Names: G-CSF

SUMMARY:
The purpose of this study is to test what effects (good and bad) a new cancer vaccine will have on participants and their cancer, when administered before and after their autologous hematopoietic cell transplant (HCT).

The name of the vaccine is called Dendritic Cell Survivin Vaccine (DC:AdmS). The vaccine is made using the participant's own blood cells. The vaccine will contain a virus called an adenovirus, similar the virus that causes the common cold. The virus has been changed so it cannot infect humans and cause infections. The vaccine will be prepared at Moffitt Cancer Center in the Cell Therapy Laboratory Facility.

DETAILED DESCRIPTION:
This study is designed to test the safety and efficacy of the survivin vaccine, as well as the biological activity. A total sample size of 30 patients will be used for the study. In the 1st stage, 10 patients will be used to evaluate the safety and futility of the vaccine. If it passes the 1st stage, investigators will enroll another 20 patients (as 2nd stage) to evaluate the efficacy. The two- stage experiment is based on Simon minmax two-stage design for efficacy. Vaccine will be administered in two stages. After the first survivin vaccination, participants will be mobilized with G-CSF and both in vivo-primed T cells and stem cells will be collected in the same apheresis (the graft). T cells and the CD34 progenitor cells will be transferred back to the participant at the time of autologous graft infusion. Participants will receive re-vaccination on, or near, day 21 after transplant.

ELIGIBILITY:
Inclusion Criteria:

Screening:

* As of protocol Version 2 there is no "screening phase".Patients previously consented to the screening phase could still be eligible for treatment if consented for treatment, based upon the updated eligibility criteria.

Treatment:

* Patients with histologically confirmed Multiple Myeloma that are being considered for high dose chemotherapy and autologous stem cell transplant.
* Patients must have a bone marrow biopsy available, or one scheduled to be performed for a clinical indication so that survivin expression could be determined (note: survivin staining in tumor need not be resulted prior to enrollment or treatment as it is obtained for correlative science).
* Patients planned for treatment with high dose melphalan and autologous hematopoietic cell transplant (HCT).
* Complete blood count (CBC) with an absolute neutrophil count (ANC) >= 1,000/uL, hemoglobin >= 8.0 g/dL and platelet count >= 50,000/uL.
* Liver enzymes: total bilirubin less than or equal to 2 mg/dL (>2 mg/dL permitted if the patient has evidence of Gilbert's disease based upon prior bilirubin elevation or genetic testing); Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) less than 1.5 X the upper limit of normal (ULN).
* Signed informed consent form in accordance with institutional and federal law policies.

Exclusion Criteria:

Treatment:

* Patients with Complete Response (CR) or stringent CR after induction therapy as defined by International Response Criteria after most recent therapy.
* Patients with progressive disease at time of transplant.
* Pregnant or lactating woman (as evaluated by serum testing within 48 hours of administration of the first vaccine in women of child bearing potential).
* HIV infection confirmed by nucleic acid tests (NAT).
* Common variable immunodeficiency.
* Active central nervous system (CNS) malignancy.
* Active bacterial, fungal or viral infection.
* Prior history of allogeneic hematopoietic cell transplantation
* Prior malignancy within 5 years of enrollment excluding non-melanoma skin cancer or cervical carcinoma after curative resection, not requiring chemotherapy.
* History of severe allergy (e.g., anaphylaxis) to any component of Prevnar or any diphtheria-toxoid containing vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Rate of Complete Response (CR) | 90 days post treatment
  Complete Response: A treatment outcome where there are ≤5% plasma cells in the bone marrow and no evidence of myeloma proteins in the serum or urine as measured by standard laboratory techniques.
Number of Participants With Treatment Emergent Adverse Events | Up to 6 months post treatment
  The safety of DC:AdmS when administered to patients with myeloma before and at day +21 after autologous hematopoietic stem cell transplant. The approach for assessing potential toxicity of survivin vaccination will focus predominantly on assessing hematopoietic reconstitution, including T cell repopulation and gastrointestinal toxicity. Investigators will also monitor for autoimmune disorders involving other tissues where survivin expression has been demonstrated: these include keratinocytes and melanocytes, myocardium, liver, breast, and brain. The most sensitive test to assess the potential toxicity of survivin vaccination on hematopoietic function is the time of neutrophil repopulation after autologous stem cell transplant (ASCT). Beginning on day of ASCT, participants will be monitored daily for engraftment, defined by an absolute neutrophil count of 500 cells per microliter that is sustained for at least 3 days.

SECONDARY OUTCOMES:
Number of Participants With Improved Immunologic Response | 180 days (6 months) post vaccination
  The ability of DC:AdmS to induce T cell immune responses against survivin when administered to patients with myeloma before and at day +21 after autologous hematopoietic stem cell transplant.
  Immunologic responses: be measured at baseline prior to the first vaccination (i.e., baseline), after stem cell mobilization and collection (i.e., pre-transplant), and post-transplant at day +60, +90, and +180. Each time 100 cc of peripheral blood will be collected. Immune response evaluations will consist of the following: Determination of the survivin specific T cell frequency using limiting dilution analysis and freely available online software; Analysis of Interferon-γ producing T cells in ELISPOT assays in response to DC loaded survivin peptide pool; Measurement of anti-pneumococcal immunoglobulin G (IgG) antibody titers and T cell responses against cross-reacting material (CRM) adjuvant; Evaluation of immunomodulatory phenotypes by T cell subsets before and after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Locke, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Freeman CL, Atkins R, Varadarajan I, Menges M, Edelman J, Baz R, Brayer J, Castaneda Puglianini O, Ochoa-Bayona JL, Nishihori T, Shain KH, Shah B, Chen DT, Kelley L, Coppola D, Alsina M, Antonia S, Anasetti C, Locke FL. Survivin Dendritic Cell Vaccine Safely Induces Immune Responses and Is Associated with Durable Disease Control after Autologous Transplant in Patients with Myeloma. Clin Cancer Res. 2023 Nov 14;29(22):4575-4585. doi: 10.1158/1078-0432.CCR-22-3987. PMID 37735756
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/